CLINICAL TRIAL: NCT05167630
Title: Prognosis Factors in Patients With Primary Central Nervous System Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Mingzhi Zhang, Dr., Zhengzhou University
Other Study IDs: hnslblzlzx20211001
Record Dates: First submitted 2021-12-12; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: PCNSL; Survival Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: prognostic marker — prognostic marker

SUMMARY:
Primary central nervous system lymphoma (PCNSL) is a rare extranodal non-hodgkin's lymphoma confined to the central nervous system. It accounts for about 4% of all intracranial tumors and 4% to 6% of all non-Hodgkin's lymphomas . Among them, the most common type is diffuse large B cell lymphoma (DLBCL), accounting for about 95% of all cases. High dose methotrexate (HD-MTX) based chemotherapy can improve the prognosis of patients, but only 30% to 40% of patients can achieve sustained remission, and the overall prognosis is very poor[4, 6]. Currently, the International Extranodal Lymphoma Study Group (IESLG) prognostic scoring system and the Memorial Sloan Kettering Cancer Center (MSKCC) prognostic index are widely used to evaluate the prognosis in patients with PCNSL. However, IESLG model has some limitations such as the relatively small number of patients and short follow-up period. MSKCC model may have an inherent selection bias because retrospective data were collected from a single large institution. Therefore, there is a urgent need to identify novel indicators for prognosis evaluation and risk stratification in PCNSL patients.

ELIGIBILITY:
Inclusion Criteria:

(i)The pathological biopsy and immunohistochemistry diagnosis were PCNSL according to WHO diagnostic criteria for PCNSL in 2016. (ii) No treatment has been received. (iii)There were no diseases with malignant tumor, serious infection, other blood system diseases, immune system diseases and other conditions which may have great influence on peripheral blood lymphocyte count. (iv) The clinical data were complete.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical data of PCNSL patients were collected retrospectively, such as sex, age, physical state (ECOG score), cell source classification, number of lesions, whether the lesions involved deep structure, etc. The data of laboratory examination include the protein content in cerebrospinal fluid, lactate dehydrogenase (LDH), β2- macroglobulin (β2-MG), IESLG score, ALC and Ki-67.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-09-01 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival | from September 1, 2013 to June 1, 2020
  from the date of diagnosis to death from any cause or to the date of last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Zhengzhou university, Zhengzhou, Henan, China